CLINICAL TRIAL: NCT01544478
Title: A Phase IV Open-Label, Descriptive Study to Evaluate the Safety and Effectiveness on the Incidence of HPV 6, 11, 16 and 18 Related CIN 2/3 or Worse of the Quadrivalent HPV (Types 6, 11, 16, 18) L1 Virus-Like Particle (VLP) Vaccine in 16- to 26-Year-Old Japanese Women
Brief Title: V501 Safety and Efficacy Study in Japanese Women Aged 16 to 26 Years (V501-110)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V501-110; 132247 (Registry Identifier: Japic-CTI); 2015-002932-42 (EudraCT Number)
Record Dates: First submitted 2012-02-29; First posted 2012-03-06 (Estimated); Results first posted 2017-07-07 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Cervical Cancer; Cervical Intraepithelial Neoplasia; Adenocarcinoma in Situ
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia; Adenocarcinoma in Situ | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- V501 (Experimental): Participants received a 0.5-mL vaccination of V501 by intramuscular injection on Day 1, Month 2, and Month 6
  Interventions: Biological: V501

INTERVENTIONS:
Biological: V501 — HPV types 6, 11, 16, and 18 vaccine 0.5 mL by intramuscular injection at Day 1, Month 2, and Month 6
  Other Names: Gardasil™

SUMMARY:
This study evaluated the long-term safety of quadrivalent Human Papillomavirus (HPV) types 6, 11, 16, 18 vaccine and its effectiveness in the prevention of cervical intraepithelial neoplasia (CIN), adenocarcinoma in situ, and cervical cancer related to HPV in Japanese women.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese females
* Not pregnant at Screening and agree to use effective contraception through Month 7 of the study
* Lifetime history of 0 to 4 male or female sexual partners
* No oral temperature ≥37.5 centigrade within 24 hours prior to injection

Exclusion Criteria:

* Received a marketed HPV vaccine
* Prior abnormal Papanicolaou smear (PAP) or biopsy showing CIN
* Known history of positive test for HPV
* Known history of genital warts
* Received immune globulin or blood products within 6 months prior to first injection or plan to receive any through Month 7 of the study
* History of splenectomy, known immune disorders, or receiving immunosuppressives
* Immunocompromised or diagnosed as having human immunodeficiency virus (HIV)

Ages: 16 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1030 (Actual)
Dates: Start 2011-11-25 (Actual); Primary Completion 2016-08-27 (Actual); Study Completion 2016-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Sakamoto M, Miyagi E, Sumi Y, Aisaka K, Kuno N, Nagano H, Asahara S, Han SR, Wakana A, Murata S, Sawata M, Tanaka Y. Effectiveness on high-grade cervical abnormalities and long-term safety of the quadrivalent human papillomavirus vaccine in Japanese women. J Infect Chemother. 2019 Jul;25(7):520-525. doi: 10.1016/j.jiac.2019.02.012. Epub 2019 Mar 15. PMID 30879979

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1036 participants were screened and 1030 were enrolled in the study.
Period: Overall Study
Arm/Group | V501
Started | 1030
Vaccination 1 | 1030
Vaccination 2 | 1026
Vaccination 3 | 1019
Completed | 912
Not Completed | 118
Not completed — Adverse Event | 1
Not completed — Death | 1
Not completed — Lost to Follow-up | 48
Not completed — Physician Decision | 15
Not completed — Pregnancy | 1
Not completed — Withdrawal by Subject | 52

BASELINE CHARACTERISTICS:
Arm/Group | V501
Number analyzed (Participants) | 1030
Age, Continuous [Mean (Standard Deviation); unit: Years] | 22.9 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1030
  Male | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 1030

OUTCOME MEASURES:

1. Primary Outcome: Combined Incidence of Cervical Intraepithelial Neoplasia (CIN) 2/3 or Worse Related to Human Papillomavirus (HPV) Type 6, 11, 16, or 18
Description: The endpoint included pathology panel consensus diagnosis of CIN 2 or 3, adenocarcinoma in situ, invasive squamous cervical carcinoma, or invasive adenocarcinoma of the cervix, and HPV type 6, 11, 16, or 18 detected in an adjacent section from the same tissue block. The point estimates and exact 95% confidence intervals for incidence rate were based on the Poisson distribution.
Time Frame: Up to Month 48
Population: The population analyzed included participants who received the full vaccination series, had at least 1 visit after Month 7, had no general protocol violations, and were seronegative at Baseline and polymerase chain reaction-negative from Baseline through Month 7 for the relevant HPV type.
Measure: Number (95% Confidence Interval); unit: Cases per 100 person-years at risk
Units Other Than Participants: Person-years at risk
Arm/Group | V501
Number analyzed (Participants) | 967
Number analyzed (Person-years at risk) | 3035
Cases per 100 person-years at risk | 0.0 [0.0 to 0.1]

ADVERSE EVENTS:
Time Frame: Up to Month 48
Description: Participants at risk included all who received at least 1 vaccination and had safety follow-up. One participant received vaccination but did not have safety follow-up.
Arm/Group | V501
Serious Adverse Events (participants affected / at risk) | 8/1029
Other Adverse Events (participants affected / at risk) | 169/1029
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V501 (N=1029)
Peritonsillitis (Infections and infestations) | 1 (1)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Abortion induced (Surgical and medical procedures) | 4 (4)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Foetal malpresentation (Pregnancy, puerperium and perinatal conditions) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V501 (N=1029)
Nasopharyngitis (Infections and infestations) | 61 (67)
Injection site pain (General disorders) | 118 (168)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.